CLINICAL TRIAL: NCT04920786
Title: A Phase 1 Double-blind, Randomized, Single Dose, Sequential Dose-escalation Study to Assess the Safety, Tolerability and Pharmacokinetics of TB006 in Healthy Subjects
Brief Title: Sequential Dose-escalation Study to Assess the Safety, Tolerability and Pharmacokinetics of TB006 in Healthy Subjects
Acronym: TB006SAD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TrueBinding, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: TB006HV1101
Record Dates: First submitted 2021-05-18; First posted 2021-06-10 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2023-02

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — TB006

STUDY DESIGN:
Intervention Model Description: Six dose groups are planned: 5 dose levels of TB006 in healthy subjects and 1 ethno-bridging group in healthy subjects of Chinese descent.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TB006 70 mg - 5000 mg IV (Experimental): TB006 infused intravenously over 1 hour
  Interventions: Drug: TB006
- Placebo (Placebo Comparator): 0.9% normal saline infused intravenously over 1 hour
  Interventions: Other: Sterile saline (Placebo)

INTERVENTIONS:
Drug: TB006 — TB006
  Arms: TB006 70 mg - 5000 mg IV
Other: Sterile saline (Placebo) — Sterile saline
  Arms: Placebo

SUMMARY:
This is a single dose, dose-escalation study to assess the safety, tolerability, pharmacokinetics and pharmacodynamics of TB006, a monoclonal antibody that will be studied as a disease modifying treatment for Alzheimer's disease.

DETAILED DESCRIPTION:
The TB006 nonclinical pharmacology program establishes its potential as a therapeutic agent for AD. Overall, the data suggest the potential for beneficial therapeutic effects of TB006 in addressing underlying pathology and ameliorating the course of AD. The preclinical safety profile of TB006 further supports the clinical investigation of TB006. This is a Phase 1 SAD study in healthy adult subjects. The study will evaluate the safety, tolerability, and PK of single doses of TB006, administered as an IV infusion over 1 hour.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers, male or female 18-55 at the time of informed consent
* In good health as determined by the principal investigator
* Body weight of ≥ 50 kg and BMI within the range 18-30 kg/m2 (inclusive).
* Chinese subjects are eligible to be included in the study if all of the following criteria apply in addition to the above: Must have been born in China, with 2 Chinese biological parents and 4 Chinese grandparents as confirmed by interview; Must have lived no more than 10 years outside of China; Must not have changed their lifestyle or habits significantly, including diet, since leaving China.

Exclusion Criteria:

* Any current history of clinically significant disease in the opinion of the investigator or receiving maintenance medications on a daily basis.
* Any active or unstable clinically significant medical or psychiatric condition as judged by the investigator.
* Smokes cigarettes or uses other nicotine-containing products (eg, snuff, nicotine patch, nicotine chewing gum, mock cigarettes, or inhalers), and has done so in the 3 months prior to screening.
* Regular alcohol consumption within 6 months prior to the study defined as: an average weekly intake of > 20 units for males or > 16 units for females. One unit is equivalent to 8 glasses of alcohol: a half pint (∼240 mL) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-05-03 (Actual); Study Completion 2022-05-03 (Actual)

PRIMARY OUTCOMES:
Number of subjects and rate of treatment-emergent adverse events, graded by CTCAE Version 5.0, by dose group and all active treatment vs. placebo | Day1-Day 75
  To measure the incidence of AEs and SAEs, clinical laboratory parameters, and vital signs until Day 75 after dosing.
To determine the single-dose PK profile of TB006 in healthy adult subjects | Through day 75
  PK parameters derived by noncompartmental analysis using the TB006 plasma concentration-time data
To determine the MTD of single doses of TB006 in healthy adult subjects | Through day 75
  Dose-response relationship of AEs and SAEs, and other safety outcomes

SECONDARY OUTCOMES:
Pharmacokinetic (PK) profile/parameters: Area under the plasma concentration versus time curve (AUC) through Day 29 | Through Day 75
  PK:AUC D0-D29
Pharmacokinetic (PK) profile/parameters: Area under the plasma concentration versus time curve (AUC) | Through Day 75
  PK: AUC D0-∞
Pharmacokinetic (PK) profile/parameters: Maximum observed plasma concentration | Through Day 75
  PK: Cmax
Pharmacokinetic (PK) profile/parameters: Time at which maximum plasma concentration occurs | Through Day 75
  PK: tmax
Pharmacokinetic (PK) profile/parameters: terminal elimination phase half life | Through Day 75
  PK: t(1/2)
Pharmacokinetic (PK) profile/parameters: total clearance | Through Day 75
  PK: CL
Pharmacokinetic (PK) profile/parameters: volume of distribution | Through Day 75
  PK: Vd
Pharmacokinetic (PK) profile/parameters: Extent of CSF distribution as estimated by TB006 CSF concentrations | Through Day 75
  PK: CSF
Safety and tolerability | Through Day 75
  Number of subjects and rate of treatment-emergent adverse events, graded by CTCAE Version 5.0, by dose group and all active treatment vs. placebo in non-Chinese healthy and Chinese healthy subjects
Anti-TB006 antibodies | Through Day 75
  Number and rate of subjects who develop anti-TB006 antibodies

CONTACTS AND LOCATIONS:
Overall Officials: George Haig, PharmD, Study Director — TrueBinding, Inc.; David Walling, MD, Principal Investigator — Collaborative Neuroscience Research
Locations (1):
- Collaborative Neuroscience Research, LLC (CNS), Long Beach, California, United States

IPD SHARING:
Plan to Share IPD: No